CLINICAL TRIAL: NCT03859050
Title: Alveolar Macrophage Programming Following Endotoxin Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-3131
Record Dates: First submitted 2019-02-14; First posted 2019-03-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-07

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LPS arm (Experimental)
  Interventions: Other: bronchoscopy with intrabronchial administration of lipopolysaccharide

INTERVENTIONS:
Other: bronchoscopy with intrabronchial administration of lipopolysaccharide — The PI will administer intrabronchial LPS into the lungs of healthy volunteers and then obtaining macrophages by bronchoalveolar lavage (BAL) 24, 48, 72, 96, or 120 hours later.

SUMMARY:
The histologic hallmarks of lung inflammation include accumulation of inflammatory cells in the airspaces and interstitium, injury to alveolar epithelial and endothelial cells, loss of epithelial-capillary integrity and accumulation of edema fluid in the interstitium and airspaces. Accordingly, for alveolar repair to occur inflammation must be halted, debris and inflammatory cells removed, injured tissue cells replaced, and capillary barrier function re-established. Macrophages are key players in all of these. Here the investigators hypothesize that resident alveolar macrophages and recruited macrophages serve completely different functions, acting independently (i.e. division of labor) yet cooperatively (synergism).

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent
2. Age 18-50

Exclusion Criteria:

1. Current or recent illness (past 2 weeks)
2. Presence or prior history of cardiac, pulmonary or systemic disease
3. Bleeding disorder, use of systemic anticoagulants or antiplatelet therapy
4. American Society of Anesthesiology (ASA) class 2 or greater
5. Immunocompromised state (HIV, immunoglobulin deficiency, systemic immunosuppressants)
6. Use of any inhaled substance, including tobacco, marijuana, e-cigarrettes, cocaine, methamphetamines, or toxic vapors in the past 3 months or greater than 10 pack-year smoking history
7. Alcohol use disorder or greater than 7 drinks/week for women or greater than 14 drinks/week for men in the past 3 months
8. Allergy or prior adverse reaction to lidocaine, midazolam or fentanyl
9. Abnormal spirometry or electrocardiogram at time of screening
10. Pregnant (based on urine pregnancy test) or breast feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Resident alveolar macrophages and recruited macrophages will be distinguished from one another using multi-parameter flow cytometry, and the relative proportions enumerated | 7 days
  Resident and recruited macrophages will be purified using fluorescence activated cell sorting (FACS) and subjected to RNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No